CLINICAL TRIAL: NCT03211221
Title: rTMS Over the Supplementary Motor Area for Treatment-resistant Obsessive-compulsive Disorder: a Multicenter, Double-blind, Controlled Trial.
Brief Title: rTMS Over the Supplementary Motor Area for Treatment-resistant Obsessive-compulsive Disorder.
Acronym: rTMSOCD
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: CNS Onlus (Other)
Collaborators: University of Florence (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Pallanti
Record Dates: First submitted 2017-07-05; First posted 2017-07-07 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: OCD; TMS
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to receive 15 sessions of active rTMS or sham rTMS over the bilateral pre-SMA with a 1:1: ratio. After the randomized phase, all patients will undergo a 4 weeks washout phase. At the end of the wash phase each patient will be classified as responder, partial responder or non-responder. After the washout phase responder patients will enter a follow-up phase up to 12 months while partial responders or non-responders in both the active and sham rTMS groups, will undergo an open phase of 15 sessions of active rTMS over the bilateral pre-SMA. Partial responders and non-responders after the randomized phase who will choose not to go into the open phase will end the study.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants, the investigators and the outcome assessor will be blind to the type of intervention (TMS or SHAM). The TMS operator will be unblinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active rTMS (Active Comparator): Active stimulation parameters will be 1-Hz, 10 seconds per train, 10 pulses per train (3 seconds inter-train interval) for a total of 160 trains (1600 pulses/session) at 130% of resting motor threshold (MT) (using the lowest value of the dominant hemisphere), once a day, 5 day/week, for 3 weeks. The coil will be positioned over the pre-SMA, targeted using the International 10-20 EEG System. Pre-SMA is defined at 15% of the distance between inion and nasion anterior to Cz (vertex) on the sagittal midline. The coil will be placed with the handle along the sagittal midline, pointing towards the occiput to stimulate bilaterally and simultaneously the pre-SMA.
  Interventions: Device: rTMS (repetitive transcranial magnetic stimulation)
- Sham rTMS (Placebo Comparator): Sham TMS will be administered by tilting the coil 90° off the scalp, with one wing of the coil touching the scalp. This sham-TMS approach produces a clicking sound that is very similar to an active TMS pulse and induces a voltage in the brain that is more than 75% lower than active TMS.
  Interventions: Device: rTMS (repetitive transcranial magnetic stimulation)

INTERVENTIONS:
Device: rTMS (repetitive transcranial magnetic stimulation) — rTMS is a non-invasive neuromodulation technique that is able to modulate cortical and subcortical function with the use of rapidly changing electromagnetic fields generated by a coil placed over the scalp (George and Post, 2011). Depending on the parameters of stimulation, rTMS can either decrease or increase cortical excitability in relatively focal areas, with frequencies < or = 1 Hz (low frequency rTMS or LF-rTMS) being usually inhibitory and higher frequencies (> or = 5 Hz; high frequency rTMS or HF-rTMS) being usually excitatory (Rosa and Lisanby, 2012). Moreover, rTMS has proven to have long-lasting effects on brain neuroplasticity through different mechanisms (e.g. by inducing long-term potentiation, increasing several neurotrophic factors etc.) (Chervyakov et al., 2015).

SUMMARY:
The aim of this study is to investigate the effectiveness of low-frequency (1Hz) rTMS (repetitive transcranial magnetic stimulation) over the pre-SMA (pre-supplementary motor area) in a sample of treatment-resistant OCD patients in a multicenter, controlled design.

DETAILED DESCRIPTION:
N consecutive treatment-resistant OCD outpatients, fulfilling all the inclusion criteria, will be recruited by each center involved in the study.

To be included in the study all the patients must be aged between 18 and 65 yy and have to meet DSM-5 criteria for OCD with a Y-BOCS total score > or = 20 and a history of treatment-resistant OCD, established by a trained psychiatrist with extensive expertise in the OCD field. Treatment-resistance is defined as non-response (less than 25% reduction of the Y-BOCS score) after at least one SRIs trials (clomipramine, fluoxetine, sertraline, paroxetine, fluvoxamine, citalopram, escitalopram) at the maximum tolerable dose for at least 12 weeks. Potential patients with any of the following conditions will be excluded: 1) any additional current psychiatric comorbidity, except for mild depressive and anxious symptoms or tics; 2) a lifetime DSM-5 diagnosis of schizophrenia or other psychotic syndromes, substance dependence or substance abuse, including alcohol, bipolar I or II disorder, mental disorder due to a general medical condition; 3) serious suicide risk; 4) episodic OCD; 5) illness duration less than two years; 6) hospitalization in the last 6 months; 7) refractory OCD (defined as non response to two SRIs trials, one antidopaminergic augmentation and at least one CBT with ERP trial); 8) patient who did not response to a previous ECT trial; 9) the inability to receive rTMS because of metallic implants, or history of seizures (personal or family history of seizure in first degree relatives); 10) any major medical disease; 11) pregnancy or nursing of an infant; 12) the inability or refusal to provide written informed consent.

No psychotherapy and/or pharmacological treatments changes will be allowed during the study period. Pharmacologically treated patients should be on constant medications for at least 6 weeks before entering the study.

Female patients included in the study will not be required to adopt contraceptive measures.

Patients with prior TMS exposure will be excluded in order to reduce the risk of unblinding.

Design of the Study Patients will be randomized to receive 15 sessions of active rTMS or sham rTMS over the bilateral pre-SMA with a 1:1: ratio. After the randomized phase, all patients will undergo a 4 weeks washout phase. During the wash out phase each patients will be re-assessed every two weeks in order to detect long-lasting rTMS effects. At the end of the wash phase each patient will be classified as responder, partial responder or non-responder. After the washout phase responder patients will enter a follow-up phase up to 12 months while partial responders or non-responders in both the active and sham rTMS groups, will undergo an open phase of 15 sessions of active rTMS over the bilateral pre-SMA. After the open rTMS phase, all patients will undergo a 4 weeks washout phase. During the wash out phase each patients will be re-assessed every two weeks in order to detect long-lasting rTMS effects. Responder patients will then continue in the follow-up phase, while non-responder or partial responders will leave the study.

Partial responders and non-responders after the randomized phase who will choose not to go into the open phase will end the study.

Study flow-chart

Active rTMS procedures Active rTMS will be administered with Magventure, Medtronic, Magandmore, Magstim, Neuronetics TMS devices using a vacuum cooled 70-mm figure-of-eight coil. Stimulation parameters will be 1-Hz, 10 seconds per train, 10 pulses per train (3 seconds inter-train interval) for a total of 160 trains (1600 pulses/session) at 130% of resting motor threshold (MT) (using the lowest value of the dominant hemisphere), once a day, 5 day/week, for 3 weeks. The coil will be positioned over the pre-SMA, targeted using the International 10-20 EEG System (Choi et al. 2006). Pre-SMA is defined at 15% of the distance between inion and nasion anterior to Cz (vertex) on the sagittal midline. The coil will be placed with the handle along the sagittal midline, pointing towards the occiput to stimulate bilaterally and simultaneously the pre-SMA.

Sham rTMS procedures Sham TMS will be administered by tilting the coil 90° off the scalp, with one wing of the coil touching the scalp (Lisamby et al., 2001). This sham-TMS approach produces a clicking sound that is very similar to an active TMS pulse and induces a voltage in the brain that is more than 75% lower than active TMS (Lisanby et al., 2001).

Motor Threshold Resting MT will be defined as the minimum magnetic flux needed to elicit a threshold EMG response (50 mV in peak-to-peak amplitude) in a resting target muscle (abductor pollicis brevis) in 5/10 trials using single-pulse TMS administered to the contralateral primary motor cortex. The motor threshold will be re-assessed every session before starting the rTMS treatment.

Side-effect ratings Before and after each session patients were asked by a blinded assessor a series of questions in a structured form in order to rate TMS side-effects. For this purpose the investigators will use the Monitoring of Side Effects Scale (MOSES).

Clinical assessment After a screening visit, the patients fulfilling the inclusion criteria will be assessed before entry the study with a comprehensive clinical interview (age, sex, education, OCD onset, OCD subtype, duration of the illness, history of past or current TICs, previews pharmacological and psychotherapeutic treatments, treatment resistance, lifetime comorbidities) and a psychometric assessment including the following tools: The SCID-5 CV (Structured Clinical Interview for DSM-5 Disorders-Clinician Version), the Yale-Brown Obsessive-Compulsive Scale (Y-BOCS), the Y-BOCS-SC (symptoms checklist) (Goodman et al., 1989a,b), the Hamilton Anxiety rating Scale (HAM-A) (Hamilton, 1959), the Hamilton Depression Rating Scale (HAM-D-17 itemes) (Hamilton, 1967) and the Clinical Global Impression Scale (CGI) (Guy, 2000).

Before starting the rTMS procedures and after 10 and 15 sessions all patients will be assessed by a blinded assessor with the following psychometric scale: Y-BOCS, HAM-D, HAM-A, CGI-S and the CGI-I. During the washput phase each patient will be re-assessed at week 2 and 4 with the Y-BOCS, HAM-D, HAM-A, CGI-S and the CGI-I.

Patients entering the open phase will be assessed after 10 and 15 sessions and at week 2 and 4 of the second washout phase with the Y-BOCS, HAM-D, HAM-A, CGI-S and the CGI-I.

Standard criteria for the treatment outcome will be included in the trial: response (>35% improvement in baseline Y-BOCS scores and a CGI-I of 1 or 2), partial response (≥ 25% improvement in baseline Y-BOCS scores), and non-response (<25% improvement in baseline Y-BOCS scores).

The end-point assessment will be repeated at 3, 6, 9 and 12 months follow-up visits after the last rTMS session in an open design.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 65 yy
* DSM-5 criteria for OCD
* Y-BOCS total score > or = 20
* History of treatment-resistant OCD, established by a trained psychiatrist with extensive expertise in the OCD field. Treatment-resistance is defined as non-response (less than 25% reduction of the Y-BOCS score) after at least one SRIs trials (clomipramine, fluoxetine, sertraline, paroxetine, fluvoxamine, citalopram, escitalopram) at the maximum tolerable dose for at least 12 weeks.

Exclusion Criteria:

* any additional current psychiatric comorbidity, except for mild depressive and anxious symptoms or tics;
* a lifetime DSM-5 diagnosis of schizophrenia or other psychotic syndromes, substance dependence or substance abuse, including alcohol, bipolar I or II disorder, mental disorder due to a general medical condition;
* serious suicide risk;
* episodic OCD;
* illness duration less than two years
* hospitalization in the last 6 months;
* refractory OCD (defined as non response to two SRIs trials, one antidopaminergic augmentation and at least one CBT with ERP trial);
* patient who did not response to a previous ECT trial;
* the inability to receive rTMS because of metallic implants, or history of seizures (personal or family history of seizure in first degree relatives);
* any major medical disease;
* pregnancy or nursing of an infant;
* the inability or refusal to provide written informed consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
rTMS effects on OC symptoms | end of the study
  Standard criteria for the treatment outcome will be included in the trial: response (>35% improvement in baseline Y-BOCS scores and a CGI-I of 1 or 2), partial response (≥ 25% improvement in baseline Y-BOCS scores), and non-response (<25% improvement in baseline Y-BOCS scores).

CONTACTS AND LOCATIONS:
Locations (1):
- Stefano Pallanti, Florence, I, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Berlim MT, Neufeld NH, Van den Eynde F. Repetitive transcranial magnetic stimulation (rTMS) for obsessive-compulsive disorder (OCD): an exploratory meta-analysis of randomized and sham-controlled trials. J Psychiatr Res. 2013 Aug;47(8):999-1006. doi: 10.1016/j.jpsychires.2013.03.022. Epub 2013 Apr 21. PMID 23615189
- [Background] Gomes PV, Brasil-Neto JP, Allam N, Rodrigues de Souza E. A randomized, double-blind trial of repetitive transcranial magnetic stimulation in obsessive-compulsive disorder with three-month follow-up. J Neuropsychiatry Clin Neurosci. 2012 Fall;24(4):437-43. doi: 10.1176/appi.neuropsych.11100242. PMID 23224449
- [Background] Mantovani A, Simpson HB, Fallon BA, Rossi S, Lisanby SH. Randomized sham-controlled trial of repetitive transcranial magnetic stimulation in treatment-resistant obsessive-compulsive disorder. Int J Neuropsychopharmacol. 2010 Mar;13(2):217-27. doi: 10.1017/S1461145709990435. Epub 2009 Aug 20. PMID 19691873